CLINICAL TRIAL: NCT04955379
Title: An Exploratory Study in Healthy Pediatric Volunteers to Evaluate the Performance of a Handheld Device Compared With Standard Eye Care Diagnostic Device in Measuring Ophthalmic Refraction
Brief Title: Study in Pediatric Volunteers of a Handheld Device Versus a Standard Diagnostic Device in Ophthalmic Refraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EyeQue Corp. (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EYEQUE-005
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Refractive Errors; Accomodation; Diagnostic Self Evaluation
Keywords: Refraction; Telehealth; Vision; Accommodation
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Measurements (Other): Subjects will be tested with the Autorefractor and the EQ103 device
  Interventions: Device: EQ103

INTERVENTIONS:
Device: EQ103 — Ophthalmic Refractometer with a measurement and background channel

SUMMARY:
This study is exploratory and examines whether the refraction results obtained from a novel optical device yields results similar to the ophthalmic refraction measurements obtained from an autorefractor in children.

DETAILED DESCRIPTION:
This study is exploratory and examines whether the refraction results obtained from a novel optical device yields results similar to the ophthalmic refraction measurements obtained from an autorefractor in the age stratum of 6 through 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages ≥6 y.o. and <18 y.o.
* Binocular vision
* Parent(s) or Guardian(s) willing and able to give informed consent on behalf of the subject.
* Subject able to follow all study procedures and requirements

Exclusion Criteria:

* Spherical correction > +8 or < -10
* Using anticholinergic medications (including first-generation antihistamines) or other medications known to affect visual acuity within the greater of 3 days or 5 half-lives prior to enrolling in this study.
* Using an investigational drug or approved therapy for investigational use within the greater of 3 days or 5 half-lives prior to enrolling in this study.
* Has initiated any new medication in the past 2 weeks that, in the best medical judgment of the investigator, would impact their participation in the study or ability to use the EyeQue EQ103 device,
* Any self/caregiver-reported mental illness or condition of the subject, including but not limited to claustrophobia, fear of simulators, nyctophobia.
* Any self/caregiver-reported neurological diseases of the subject, including but not limited to: epilepsy, nystagmus.
* Any self/caregiver-reported glaucoma diagnosis of the subject.
* Eye disease, including but not limited to:

  * Cataracts
  * Macular degeneration
  * Eye infection (by self-report or observation)
  * Keratoconus
  * Diabetic neuropathy/retinopathy
  * Cytomegalovirus retinitis
  * Color blindness (any color deficiency)
  * Diabetic macular edema
  * Amblyopia
  * Chronic or acute uveitis
  * Strabismus
  * Astigmatism > 3 diopters
  * Macular hole
* Lack physical dexterity to properly operate the EyeQue device.
* Lack the ability to follow instruction.
* Lack binocular vision.
* Are colorblind.
* Had eye surgery within the last 12 months.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Tendency of, or achieving, statistical equivalence of refraction measurements EQ103 (non-cycloplegic) compared with autorefractor (non-cycloplegic) | Day 1
  Tendency of, or achieving, statistical equivalence of refraction measurements EQ103 (non-cycloplegic) compared with autorefractor (non-cycloplegic)

SECONDARY OUTCOMES:
EyeQue EQ103 (non-cycloplegic) and the autorefractor (cycloplegic) assessed by refractive error measured by each device analyzed by age-strata. | Day 1 and 14
  EyeQue EQ103 (non-cycloplegic) and the autorefractor (cycloplegic) assessed by refractive error measured by each device analyzed in the following age-strata.
  Age Groups
  * 6 to 12 y.o. >12 to <18 y.o.
EyeQue EQ103 (non-cycloplegic) and the autorefractor (cycloplegic) assessed by refractive error measured by each device analyzed by age-strata. | Day 1 and 14
  EyeQue EQ103 (non-cycloplegic) and the autorefractor (cycloplegic) assessed by refractive error measured by each device analyzed in the following age-strata.
  Age Group
  * 6 to 12 y.o.
EQ103 without cycloplegia will be compared to EQ103 with cycloplegia by younger age-strata. | Day 1 and 14
  EQ103 without cycloplegia will be compared to EQ103 with cycloplegia in the following age-strata.
  Age Group
  * 6 to 12 y.o.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Sapiens, PhD, Study Director — Sponsor GmbH
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No